CLINICAL TRIAL: NCT06607458
Title: An Open-label, Randomized, Multi-Center Study to Evaluate the Efficacy and Safety of Induction Treatment With Melphalan/HDS Followed by Consolidation Treatment With Trifluridine-Tipiracil Plus Bevacizumab Versus Trifluridine-Tipiracil Plus Bevacizumab Alone in Patients With Refractory Metastatic Colorectal Cancer With Liver Dominant Disease
Brief Title: Evaluation of the Safety and Efficacy of Treatment w/High Dose Melphalan Given Directly Into the Liver Followed by Treatment w/Approved Cancer Treatment or Approved Cancer Treatment Alone in Patients w/ Metastatic Colorectal Cancer w/Liver Dominant Disease
Acronym: DEL-LIVER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHP-CRC-201
Record Dates: First submitted 2024-09-14; First posted 2024-09-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: melphalan/HDS; melphalan/hepatic delivery system; trifluridine-tipiracil; trifluridine-tipiracil (FTD-TPI); trifluridine-tipiracil (FTD-TPI) plus bevacizumab; trifluridine-tipiracil plus bevacizumab; hepatic delivery system; melphalan; liver dominant disease; colorectal cancer; metastatic colorectal cancer; refractory metastatic colorectal cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melphalan/HDS followed by Consolidation Treatment with Trifluridine-tipiracil plus Bevacizumab (Experimental): Melphalan/HDS is given as an infusion of Melphalan into the hepatic artery under general anesthesia. This treatment is administered twice, 8 weeks apart. Following 2 treatments with Melphalan/HDS, Trifluridine-tipiracil is given 35 mg/m2 up to a maximum of 80 mg per dose orally twice daily with food on Days 1 through 5 and Days 8 through 12 of each 28-day cycle; and intravenous (IV) bevacizumab 5 mg/kg body weight on Days 1 and 15 of each 28-day cycle until disease progression or unacceptable toxicity
  Interventions: Drug: Melphalan/HDS Followed by Consolidation Treatment with Trifluridine-tipiracil plus Bevacizumab
- Trifluridine-tipiracil plus Bevacizumab Alone (Active Comparator): Trifluridine-tipiracil plus Bevacizumab is the standard of care for patients with metastatic colorectal cancer. Trifluridine-tipiracil is given 35 mg/m2 up to a maximum of 80 mg per dose orally twice daily with food on Days 1 through 5 and Days 8 through 12 of each 28-day cycle; and intravenous (IV) bevacizumab 5 mg/kg body weight on Days 1 and 15 of each 28-day cycle until disease progression or unacceptable toxicity
  Interventions: Drug: Trifluridine-tipiracil plus Bevacizumab Alone

INTERVENTIONS:
Drug: Melphalan/HDS Followed by Consolidation Treatment with Trifluridine-tipiracil plus Bevacizumab — Trifluridine-tipiracil plus Bevacizumab Alone
  Other Names: Melphalan; HDS; Trifluridine-tipiracil plus Bevacizumab; Trifluridine-tipiracil; Melphalan/HDS
  Arms: Melphalan/HDS followed by Consolidation Treatment with Trifluridine-tipiracil plus Bevacizumab
Drug: Trifluridine-tipiracil plus Bevacizumab Alone — Trifluridine-tipiracil plus Bevacizumab Alone
  Other Names: Trifluridine-tipiracil; Bevacizumab
  Arms: Trifluridine-tipiracil plus Bevacizumab Alone

SUMMARY:
The goal of this clinical trial is to learn if using a liver-directed therapy with high dose chemotherapy followed by approved cancer treatment to treat patients with colorectal cancer that has spread to the liver is safe and tolerable. The clinical trial will also learn if the liver-directed therapy with high dose chemotherapy works on the disease in the liver. Investigators will compare the use of the liver-directed therapy with high dose chemotherapy followed by approved cancer treatment or approved cancer treatment alone.

Participants will:

* Undergo up to two liver-directed therapy with high dose chemotherapy procedures followed by approved cancer treatment or take approved cancer treatment alone
* Visit clinic at least every two weeks for checkups and tests
* Complete scans approximately every two months

DETAILED DESCRIPTION:
This is an open-label, randomized, multi-center study in which patients with liver dominant refractory mCRC will be randomized 2:1 to receive melphalan/HDS (2 cycles) followed by trifluridine-tipiracil plus bevacizumab treatment (Arm A) or trifluridine-tipiracil plus bevacizumab alone (Arm B).

Approximately 90 patients will be randomized 2:1 to the two treatment arms (Arm A, n=60; Arm B, n=30). Patients will receive one of the following treatments:

* Arm A: Patients will be treated with melphalan/HDS 3.0 mg/kg ideal body weight (IBW) for two treatment cycles. The second melphalan/HDS treatment will be administered 8 weeks after the first treatment with an acceptable delay of up to 2 weeks (10 weeks total) to allow for recovery of melphalan-related toxicity, if needed. Tumor response will be assessed every 8 weeks (± 3 days) during melphalan/HDS treatment, i.e., prior to Cycle 2 of melphalan/HDS and prior to the start of trifluridine-tipiracil plus bevacizumab treatment.
* Arm B: Patients will be treated with standard regimen of trifluridine-tipiracil and bevacizumab.

In both treatment arms, treatment with trifluridine-tipiracil plus bevacizumab will continue until disease progression, death, intolerable adverse events, consent withdrawal, principal investigator decision, or termination of study by Sponsor.

Cross-over: There will be no cross-over between the two arms of the study. Efficacy and Safety Assessment: Evaluation of tumor response will be determined by the local principal investigator using RECIST 1.1 criteria. Tumor response evaluation and patient management will be according to the principal investigator assessment of images and patients' clinical needs. Patients with progressive disease (PD) will be discontinued from study treatment and will be followed for survival until withdrawal of consent or death.

Study treatment will be discontinued if recovery from treatment related toxicity requires more than 2 weeks from the end of the treatment cycle during melphalan/HDS cycles (Arm A only), or more than a 28-day delay in the start of the next cycle of trifluridine-tipiracil plus bevacizumab; the end of treatment (EOT) visit will be conducted at that time or within 4 weeks.

Safety will be monitored continuously by documentation of AEs, SAEs, clinical laboratory measurements, vital signs, and physical examination.

Data Safety Monitoring Board (DSMB): A DSMB including independent (non-investigator) clinicians will oversee the emerging patient safety profile during the study. The DSMB will review study data on a regular basis according to the DSMB Charter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of metastatic colorectal cancer and histologically or cytologically proven CRC metastases that occupy 50% or less of the liver parenchyma.
* Patient has liver-dominant metastatic disease. Liver-dominant is defined as the majority of total tumor burden is located in the liver, and the liver lesions are not resectable or treatable with ablation or are associated with extrahepatic disease that makes surgical intervention non-curative.
* Disease in the liver must be measurable (per RECIST v.1.1 guidelines) by computed tomography (CT) and/or magnetic resonance imaging (MRI).
* If there is evidence of extrahepatic metastatic disease, it is limited, and the life-threatening component of disease is in the liver. Limited extrahepatic disease is defined in this protocol as follows: up to 5 tumor lesions in the lung with longest diameter not greater than 2 cm and/or up to 5 lymph nodes that measure 2 cm or less per lesion; solitary lesions definitively treated with no sign of progression in the last 6 months.
* Scans used to determine eligibility (CT scan of the chest/abdomen/pelvis and MRI of the liver) must be performed within 28 days prior to randomization.
* Previous treatment and progressed on or following, or intolerant to, fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and/or an anti-EGFR therapy if RAS wild-type.
* ECOG PS of 0-1 within 14 days prior to randomization.

Exclusion Criteria:

* Child-Pugh Class B or C cirrhosis or evidence of clinically significant portal hypertension by history, endoscopy, or radiologic studies (large abdominal varices, prior history of varices by endoscopy).
* New York Heart Association functional classification II, III or IV or active cardiac condition(s), including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias, or severe valvular disease that create(s) undue risks of undergoing general anesthesia.
* History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia.
* History of bleeding disorders, presence of brain metastases, or other intracranial abnormalities found on baseline radiologic imaging that would put them at risk for bleeding with anti-coagulation.
* Known varices at risk of bleeding, including medium or large esophageal or gastric varices, active peptic ulcer, or history of recent hemoptysis.
* Active second malignancy, or has history of recently definitively treated invasive cancer in the past 2 years prior to enrolment with the exception of non-melanoma skin cancer.
* Peritoneal lesions or large abdominal masses.
* Use of immunosuppressive drugs.
* Inability to temporarily stop chronic anti-coagulation therapy.
* Active bacterial infections with systemic manifestations.
* Active viral infection, including Hepatitis B and Hepatitis C infection. NOTE: Patients with anti-hepatitis B core antibody (HBc) positive, or hepatitis B surface antigen (HBsAg) but DNA negative are allowed exception(s).
* Severe allergic reaction to iodine contrast that cannot be controlled by premedication with antihistamines and steroids.
* History of or known hypersensitivity to melphalan or the components of the melphalan/HDS system.
* History of known hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia.
* Uncontrolled endocrine disorder including diabetes mellitus, hypothyroidism, or hyperthyroidism.
* Received anti-cancer therapy including radiotherapy or investigational agent for any indication ≤ 30 days prior to randomization
* Previous treatment with trifluridine-tipiracil.
* History of allergic reactions attributed to compounds of similar composition to trifluridine/tipiracil or any of its excipients.
* Hereditary problems of galactose intolerance, total lactase deficiency or glucosegalactose malabsorption.
* History of allergic reactions or hypersensitivity to bevacizumab or any of its excipients.
* History of hypersensitivity to Chinese Hamster Ovary cell products or other recombinant human or humanized antibodies.
* Contraindications to bevacizumab, including uncontrolled hypertension, history of active fistula or bowel perforation (unless in the setting of a resected primary), history of CVA or arterial thrombotic event in the last 1 year, or history of venous thrombotic event in the last 30 days.
* Evidence of hepatic vein or portal vein thrombosis
* Prior chemoembolization or radioembolization to the liver or prior hepatic arterial infusion therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
hPFS | time from randomization to the first occurrence of hepatic disease progression, assessed over 24 months
  Hepatic Progression Free Survival

SECONDARY OUTCOMES:
PFS | time from randomization to the first occurrence of progression, assessed up to 24 months
  Progression Free Survival
OS | time from randomization date to the date of death due to any cause, assessed up to 36 months
  Overall Survival
ORR | Baseline through completion of treatment, assessed up to 24 months
  Overall Response Rate complete response [CR] + partial response [PR]
hORR | assessed from Baseline until there is evidence of disease progression in the liver, assessed up to 24 months
  Hepatic Overall Response Rate
DOR | assessed from Baseline until there is evidence of disease progression, assessed up to 24 months
  Duration of Response
DCR | complete response of any duration, partial response of any duration, or stable disease for a minimum of 12 weeks from randomization date, assessed up to 24 months
  Disease Control Rate
hDOR | assessed from Baseline until there is evidence of hepatic disease progression, assessed up to 24 months
  Hepatic Duration of Response
hDCR | complete hepatic response of any duration, partial response of any duration, or stable disease for a minimum of 12 weeks from randomization date, assessed up to 24 months
  Hepatic Disease Control Rate

OTHER OUTCOMES:
Safety and Tolerability | assessed from signed informed consent form until study completion
  Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) Changes from baseline in physical examination findings, vital signs, clinical laboratory parameters, electrocardiogram (ECG) and echocardiogram (ECHO) parameters

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (6):
- United States (3):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Clinical Research Center, Fairway, Kansas
- Helios Park-Klinikum Leipzig, Leipzig, Germany
- Instiuto Europeo de Oncologia, Milan, Italy
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Delcath does not currently have a plan to share IPD